CLINICAL TRIAL: NCT00006363
Title: Phase III Randomized Study of Induction Chemotherapy With or Without MDR-Modulation With PSC-833 (NSC # 648265, IND # 41121) Followed by Cytogenetic Risk-Adapted Intensification Therapy Followed by Immunotherapy With rIL-2 (NSC # 373364, IND # 1969) vs. Observation in Previously Untreated Patients With AML < 60 Years
Brief Title: Combination Chemotherapy With or Without PSC 833, Peripheral Stem Cell Transplantation, and/or Interleukin-2 in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02824; CALGB-19808; U10CA031946 (NIH)
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Erythroid Leukemia (M6); Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monoblastic Leukemia and Acute Monocytic Leukemia (M5); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Childhood Acute Basophilic Leukemia; Childhood Acute Eosinophilic Leukemia; Childhood Acute Erythroleukemia (M6); Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Minimally Differentiated Myeloid Leukemia (M0); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monoblastic Leukemia and Acute Monocytic Leukemia (M5); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloblastic Leukemia With Maturation (M2); Childhood Acute Myeloblastic Leukemia Without Maturation (M1); Childhood Acute Myelomonocytic Leukemia (M4); Childhood Myelodysplastic Syndromes; de Novo Myelodysplastic Syndromes; Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute | interventions — Cytarabine; Daunorubicin; Etoposide; valspodar; Filgrastim; Granulocyte Colony-Stimulating Factor; Busulfan; Peripheral Blood Stem Cell Transplantation; aldesleukin; Interleukin-2; Watchful Waiting; Observation

ARMS (7):
- Induction Arm I (Experimental): Patients receive cytarabine IV continuously on days 1-7 and daunorubicin IV over 5-10 minutes followed by etoposide IV over 2 hours on days 1-3. Patients with 20% or greater bone marrow cellularity and greater than 5% leukemia blasts at the end of the first course receive a second course of cytarabine IV continuously on days 1-5 and daunorubicin IV over 5-10 minutes followed by etoposide IV over 2 hours on days 1 and 2.
  Interventions: Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Other: pharmacological study
- Induction Arm II (Experimental): Patients receive PSC 833 IV continuously on days 1-3 and cytarabine, daunorubicin, and etoposide as in arm I. Patients with 20% or greater bone marrow cellularity and greater than 5% leukemia blasts at the end of the first course receive a second course of PSC 833 IV continuously on days 1 and 2 and cytarabine, daunorubicin, and etoposide as in arm I.
  Interventions: Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: etoposide; Drug: valspodar; Other: pharmacological study
- Intensification Favorable (Experimental): Patients receive HiDAC IV over 3 hours every 12 hours on days 1, 3, and 5. Treatment repeats no earlier than 28 days after the prior course and no later than 14 days after hematopoietic recovery for two more courses.
  Interventions: Drug: cytarabine; Other: pharmacological study
- Intensification Unfavorable PBSCT Group (Experimental): Patients receive etoposide IV continuously and HiDAC IV over 2 hours every 12 hours on days 1-4. Patients also receive G-CSF SC daily beginning on day 14 and continuing until PBSC collection is completed. Patients who are not able to undergo PBSCT after HiDAC/etoposide continue treatment in the non-PBSCT group. At least 4 weeks after HiDAC/etoposide recovery, patients receive oral busulfan every 6 hours on days -7 to -4 and etoposide IV over 4 hours on day -3 prior to PBSCT. Patients receive autologous PBSC infusion on day 0. Patients also receive G-CSF SC beginning on day 0 and continuing until hematopoietic recovery.
  Interventions: Drug: cytarabine; Drug: etoposide; Biological: filgrastim; Drug: busulfan; Procedure: autologous hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Other: pharmacological study
- Intensification Unfavorable Non-PBSCT Group (Experimental): Patients receive etoposide, HiDAC, and G-CSF as in the PBSCT group. After hematopoietic recovery, patients then receive HiDAC IV over 3 hours every 12 hours on days 1, 3, and 5. Treatment repeats no earlier than 28 days after prior course and no later than 14 days after hematopoietic recovery for one more course.
  Interventions: Drug: cytarabine; Drug: etoposide; Biological: filgrastim; Other: pharmacological study
- Immunotherapy Arm I (Experimental): Patients begin therapy no later than 120 days after the first day of the last course of HiDAC treatment OR day 0 of PBSCT. Patients receive low-dose IL-2 SC on days 1-14, 19-28, 33-42, 47-56, 61-70, and 75-90. In addition, patients receive high-dose IL-2 SC on days 15-17, 29-31, 43-45, 57-59, and 71-73.
  Interventions: Biological: aldesleukin; Other: pharmacological study
- Immunotherapy Arm II (Active Comparator): Patients are observed and receive no further therapy.
  Interventions: Other: clinical observation; Other: pharmacological study

INTERVENTIONS:
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
  Arms: Induction Arm I; Induction Arm II; Intensification Favorable; Intensification Unfavorable Non-PBSCT Group; Intensification Unfavorable PBSCT Group
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; daunomycin hydrochloride; daunorubicin; RP-13057
  Arms: Induction Arm I; Induction Arm II
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Induction Arm I; Induction Arm II; Intensification Unfavorable Non-PBSCT Group; Intensification Unfavorable PBSCT Group
Drug: valspodar — Given IV
  Other Names: Amdray; PSC 833
  Arms: Induction Arm II
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
  Arms: Intensification Unfavorable Non-PBSCT Group; Intensification Unfavorable PBSCT Group
Drug: busulfan — Given orally
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
  Arms: Intensification Unfavorable PBSCT Group
Procedure: autologous hematopoietic stem cell transplantation — Undergo autologous PBSCT
  Arms: Intensification Unfavorable PBSCT Group
Procedure: peripheral blood stem cell transplantation — Undergo autologous PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
  Arms: Intensification Unfavorable PBSCT Group
Biological: aldesleukin — Given SC
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
  Arms: Immunotherapy Arm I
Other: clinical observation — Undergo clinical observation
  Other Names: observation
  Arms: Immunotherapy Arm II
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. PSC 833 may increase the effectiveness of chemotherapy by making cancer cells more sensitive to the drugs. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. This randomized phase III trial is studying giving combination chemotherapy together with PSC 833 followed by a peripheral stem cell transplant with or without interleukin-2 to see how well it works compared to combination chemotherapy alone followed by a peripheral stem cell transplant with or without interleukin-2 in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of PSC-833 (valspodar) to induction chemotherapy improves disease-free survival and overall survival for patients with acute myeloid leukemia (AML) < 60 years.

II. To determine whether post-consolidation immunotherapy with low-dose continuous/intermittent high-dose bolus subcutaneous recombinant interleukin-2 (rIL-2) (aldesleukin) improves disease-free survival and overall survival in patients with AML < 60 years in first complete remission (CR).

SECONDARY OBJECTIVES:

I. To continue to evaluate the effectiveness of three courses of high-dose ARA-C (HiDAC) (cytarabine) as curative consolidation chemotherapy in patients with core binding factor (CBF) leukemias.

II. To continue to establish the use of intensive post-remission chemotherapy with PSCT or a novel intensification sequence consisting of HiDAC/high-dose etoposide/G-CSF (filgrastim) followed by two cycles of HiDAC in patients in CR with unfavorable cytogenetics.

III. To correlate the rate of relapse and toxicity with busulfan pharmacokinetics when busulfan and etoposide are used prior to autologous stem cell transplantation for AML patients in first CR.

OUTLINE: This is a randomized, multicenter study.

INDUCTION THERAPY: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cytarabine IV continuously on days 1-7 and daunorubicin IV over 5-10 minutes followed by etoposide IV over 2 hours on days 1-3. Patients with 20% or greater bone marrow cellularity and greater than 5% leukemia blasts at the end of the first course receive a second course of cytarabine IV continuously on days 1-5 and daunorubicin IV over 5-10 minutes followed by etoposide IV over 2 hours on days 1 and 2.

ARM II: Patients receive PSC 833 IV continuously on days 1-3 and cytarabine, daunorubicin, and etoposide as in arm I. Patients with 20% or greater bone marrow cellularity and greater than 5% leukemia blasts at the end of the first course receive a second course of PSC 833 IV continuously on days 1 and 2 and cytarabine, daunorubicin, and etoposide as in arm I.

INTENSIFICATION THERAPY: Patients in complete remission receive intensification therapy. Therapy begins no earlier than 2 weeks and no later than 4 weeks after complete remission is attained. Patients are stratified according to cytogenetics (favorable [t(8;21)(q22;q22) or inv(16)(p13;q22) or t(16;16)(p13;q22)] vs unfavorable [all other karyotypes]).

FAVORABLE: Patients receive high-dose cytarabine (HiDAC) IV over 3 hours every 12 hours on days 1, 3, and 5. Treatment repeats no earlier than 28 days after the prior course and no later than 14 days after hematopoietic recovery for two more courses.

UNFAVORABLE: Patients are further divided into two groups based on ability to receive peripheral blood stem cell transplantation (PBSCT) (yes vs no).

PBSCT GROUP: Patients receive etoposide IV continuously and HiDAC IV over 2 hours every 12 hours on days 1-4. Patients also receive filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 14 and continuing until peripheral blood stem cell (PBSC) collection is completed. Patients who are not able to undergo PBSCT after HiDAC/etoposide continue treatment in the non-PBSCT group. At least 4 weeks after HiDAC/etoposide recovery, patients receive oral busulfan every 6 hours on days -7 to -4 and etoposide IV over 4 hours on day -3 prior to PBSCT. Patients receive autologous PBSC infusion on day 0. Patients also receive G-CSF SC beginning on day 0 and continuing until hematopoietic recovery.

NON-PBSCT GROUP: Patients receive etoposide, HiDAC, and G-CSF as in the PBSCT group. After hematopoietic recovery, patients then receive HiDAC IV over 3 hours every 12 hours on days 1, 3, and 5. Treatment repeats no earlier than 28 days after prior course and no later than 14 days after hematopoietic recovery for one more course.

IMMUNOTHERAPY: Patients are again randomized to 1 of 2 treatment arms.

ARM I: Patients begin therapy no later than 120 days after the first day of the last course of HiDAC treatment OR day 0 of PBSCT. Patients receive low-dose interleukin-2 (IL-2) SC on days 1-14, 19-28, 33-42, 47-56, 61-70, and 75-90. In addition, patients receive high-dose IL-2 SC on days 15-17, 29-31, 43-45, 57-59, and 71-73.

ARM II: Patients are observed and receive no further therapy.

Patients are followed at 1 month, every 2 months for 2 years, every 6 months for 2 years, and then annually for 6 years.

PROJECTED ACCRUAL: A total of 720 patients will be accrued for this study within 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal histologic diagnosis of AML (> 20% blasts in the bone marrow based on the World Health Organization [WHO] and/or French-American-British Cooperative group [FAB] classifications), excluding M3 (acute promyelocytic leukemia); patients with antecedent myelodysplasia are eligible for treatment on this trial only if there was no bone marrow biopsy showing myelodysplastic syndrome (MDS) > 3 months prior to enrollment; patients with therapy-related MDS or therapy-related AML or a chronic myeloproliferative disorder are not eligible
* No prior treatment for leukemia or myelodysplasia with four permissible exceptions:

  * Emergency leukapheresis
  * Emergency treatment for hyperleukocytosis with hydroxyurea
  * Cranial radiation therapy (RT) for central nervous system (CNS) leukostasis (one dose only)
  * Growth factor/cytokine support

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 720 (Actual)
Dates: Start 2000-11; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Up to 10 years
  An unstratified logrank test for the induction treatment comparison and a stratified logrank test for the post-remission treatment comparison will be the primary statistical methods used for treatment comparisons.
Overall survival | Up to 10 years
  An unstratified logrank test for the induction treatment comparison and a stratified logrank test for the post-remission treatment comparison will be the primary statistical methods used for treatment comparisons.

SECONDARY OUTCOMES:
Estimates of disease-free survival curves | Up to 10 years
Estimates of overall survival curves | Up to 10 years
Toxicities and adverse events assessed using National Cancer Institute (NCI) Common Toxicity Criteria (CTC) | Up to 10 years
  Will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kolitz, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States

REFERENCES:
- [Derived] Seffernick AE, Mrozek K, Nicolet D, Stone RM, Eisfeld AK, Byrd JC, Archer KJ. High-dimensional genomic feature selection with the ordered stereotype logit model. Brief Bioinform. 2022 Nov 19;23(6):bbac414. doi: 10.1093/bib/bbac414. PMID 36184192
- [Derived] Walker CJ, Kohlschmidt J, Eisfeld AK, Mrozek K, Liyanarachchi S, Song C, Nicolet D, Blachly JS, Bill M, Papaioannou D, Oakes CC, Giacopelli B, Genutis LK, Maharry SE, Orwick S, Archer KJ, Powell BL, Kolitz JE, Uy GL, Wang ES, Carroll AJ, Stone RM, Byrd JC, de la Chapelle A, Bloomfield CD. Genetic Characterization and Prognostic Relevance of Acquired Uniparental Disomies in Cytogenetically Normal Acute Myeloid Leukemia. Clin Cancer Res. 2019 Nov 1;25(21):6524-6531. doi: 10.1158/1078-0432.CCR-19-0725. Epub 2019 Aug 2. PMID 31375516
- [Derived] Kolitz JE, George SL, Marcucci G, Vij R, Powell BL, Allen SL, DeAngelo DJ, Shea TC, Stock W, Baer MR, Hars V, Maharry K, Hoke E, Vardiman JW, Bloomfield CD, Larson RA; Cancer and Leukemia Group B. P-glycoprotein inhibition using valspodar (PSC-833) does not improve outcomes for patients younger than age 60 years with newly diagnosed acute myeloid leukemia: Cancer and Leukemia Group B study 19808. Blood. 2010 Sep 2;116(9):1413-21. doi: 10.1182/blood-2009-07-229492. Epub 2010 Jun 3. PMID 20522709